CLINICAL TRIAL: NCT00714363
Title: Comparison of Laser-Assisted in Situ Keratomeleusis (LASIK) vs Sub-Bowman's Keratomileusis (SBK): Assessment of Visual Function and Patient Satisfaction
Brief Title: Comparison of LASIK and SBK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Majid Moshirfar, MD, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25514
Record Dates: First submitted 2008-07-08; First posted 2008-07-14 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2010-10

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Keratomileusis, Laser In Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): LASIK
  Interventions: Procedure: LASIK
- 2 (Active Comparator): SBK
  Interventions: Procedure: SBK

INTERVENTIONS:
Procedure: LASIK — Refractive surgery
  Arms: 1
Procedure: SBK — Refractive surgery
  Arms: 2

SUMMARY:
The objective of the study is to compare clinical outcomes from LASIK and SBK using FDA-approved laser technology on the same patient

DETAILED DESCRIPTION:
Patients undergoing bilateral refractive surgery on the same day will have one eye randomized to LASIK and the fellow eye assigned to SBK treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients deemed to be suitable candidates for bilateral LASIK surgery

Exclusion Criteria:

* Patients who desire monovision correction rather than bilateral distance correction

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-10; Primary Completion 2008-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Visual acuity | 6 months

SECONDARY OUTCOMES:
Manifest refraction | 6 months
Wavefront aberration value | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Majid Moshirfar, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, John Moran Eye Center, Salt Lake City, Utah, United States